CLINICAL TRIAL: NCT02121327
Title: Disease Management Program (DMP) Stroke Trial
Brief Title: The Effects of Disease Management Programs for Prevention of Recurrent Ischemic Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hiroshima University (Other)
Collaborators: Ministry of Health, Labour and Welfare, Japan (Other Government)
Responsible Party: Principal Investigator, Michiko Moriyama, Institute of biomedical and health sciences, Hiroshima University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 21171401
Record Dates: First submitted 2014-01-15; First posted 2014-04-23 (Estimated); Last update posted 2018-02-22 (Actual); Status verified 2018-02

CONDITIONS: Ischemic Stroke
Keywords: stroke, disease management programs, self-management
MeSH Terms: conditions — Ischemic Stroke; Stroke | interventions — Disease Management

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- usual care (Active Comparator): usual care group receive regular outpatient treatment
  Interventions: Other: usual care
- disease management (Experimental): desease management program include self management education by nurse on 6months.
  Interventions: Other: disease management; Other: usual care

INTERVENTIONS:
Other: disease management — disease management program include self management education
  Other Names: Intervention of disease management program
  Arms: disease management
Other: usual care — usual care group receive regular outpatient treatment

SUMMARY:
It has been reported that stroke is the first cause of becoming bedridden, and its cumulative recurrence rate in 5 years is approximately 35%. There is a high probability that patients reduce or discontinue medications by self-determination, leading to a high risk of stroke recurrence in these patients. Comprehensive and long-term patient educations ameliorating their self-management are important making patients possible to be managed according to the guidelines for their risk factors. Using disease management programs created for each of risk factors according to clinical practice guidelines, the influence of those programs were evaluated for the prevention of stroke recurrence in this Disease Management Program Stroke Trial.

ELIGIBILITY:
Inclusion Criteria:

* Ischemic stroke onset [including transient ischemic attack (TIA)].
* Receiving regular consultation with their primary care physician.
* modified Rankin Scale (mRS) score from 0 to 3 at discharge.

Exclusion Criteria:

* modified Rankin Scale (mRS) score 4 and over at discharge .
* Patient having severe complications and the physical symptom that the contents of the program cannot carry out.
* They had medical care in medical/nursing care institutions.
* Patients with pregnancy or under terminal care.
* Dementia (scores of ≤20/30 on the Revised Hasegawa's Dementia Scale) However, when a care-giving family member living with the patient could provide self-management, patients were included even if they had dementia.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 321 (Actual)
Dates: Start 2010-09 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Framingham Risk Score: general cardiovascular disease 10 year risk | 2.5 years
  Use score of Framingham Risk Score: general cardiovascular disease 10 year risk

SECONDARY OUTCOMES:
Cumulative incidence rate of stroke recurrence and the complication (cardiovascular disease) | 2.5 years
  Questionnaire to a patient, and checking it by a nurse
All-cause mortality | 2.5 years
  Questionnaire to a patient, and checking it by a nurse
body weight | 2.5 years
  Questionnaire to a patient
body mass index | 2.5 years
  Calculation of height and the weight of the patient
blood pressure | 2.5 years
  Questionnaire to a patient
cholesterol | 2.5 years
  total cholesterol, high-density lipoprotein cholesterol, low-density lipoprotein cholesterol, triglyceride The patient mails the copy of the blood test result
serum creatinine | 2.5 years
  The patient mails the copy of the blood test result
blood urea nitrogen | 2.5 years
  The patient mails the copy of the blood test result
glycated hemoglobin (HbA1c) | 2.5 years
  The patient mails the copy of the blood test result
blood glucose | 2.5 years
  The patient mails the copy of the blood test result
prothronbin time international rate | 2.5 years
  only as for the necessary paticipant The patient mails the copy of the blood test result
Mental Depression degree | 2.5 years
  Using score of The Center for Epidemiologic Depression Scale (CES-D)
self-efficacy degree | 2.5 years
  Using score of self-efficacy scale on health behavior in patient with chronic disease
Qiality of Life (QOL) degree | 2.5 years
  Using score of MOS 36-item short form (SF-36)
Evaluated subject frequency of checking blood pressure | 2.5 years
  Questionnaire to a patient
Evaluated subject frequency of taking medicine | 2.5 years
  Questionnaire to a patient
Evaluated subject frequency of keeping the prescribed diet | 2.5 years
  Questionnaire to a patient
Evaluated subject frequency of exercising | 2.5 years
  Questionnaire to a patient

CONTACTS AND LOCATIONS:
Overall Officials: Michiko Moriyama, RN, PhD., Principal Investigator — Hiroshima University
Locations (1):
- Hiroshima University, Hiroshima, Hiroshima, Japan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Crocker TF, Brown L, Lam N, Wray F, Knapp P, Forster A. Information provision for stroke survivors and their carers. Cochrane Database Syst Rev. 2021 Nov 23;11(11):CD001919. doi: 10.1002/14651858.CD001919.pub4. PMID 34813082
- [Derived] Fukuoka Y, Hosomi N, Hyakuta T, Omori T, Ito Y, Uemura J, Yagita Y, Kimura K, Matsumoto M, Moriyama M; for DMP Stroke Trial Investigators. Effects of a Disease Management Program for Preventing Recurrent Ischemic Stroke. Stroke. 2019 Mar;50(3):705-712. doi: 10.1161/STROKEAHA.118.020888. PMID 30802185